CLINICAL TRIAL: NCT07176988
Title: Deconstructing Voice Therapy: Towards Enhanced Communication Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Amanda Gillespie, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00009121; 1R01DC022026-01A1 (NIH)
Record Dates: First submitted 2025-08-18; First posted 2025-09-16 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Dysphonia; Primary Muscle Tension Dysphonia (MTD)
Keywords: Conversation Training Therapy; Hierarchical Conversation Training Therapy; primary muscle tension dysphonia; benign vocal fold lesions
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned based on a stratified block randomization based on diagnosis (MTD, lesions), severity (mild, moderate, severe), and sex
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-Hierarchical Conversation Training Therapy (CTT) (Experimental)
  Interventions: Other: Non Hierarchical method
- Hierarchical Conversation Training Therapy (CTT-H) (Experimental)
  Interventions: Other: Hierarchical method

INTERVENTIONS:
Other: Hierarchical method — Participants in the hierarchical version of Conversation Training Therapy (CTTH) will receive four weekly sessions of voice therapy. This approach gradually increases the difficulty of speaking tasks-from simple sounds to full conversations-based on the participant's progress. The therapy begins with basic awareness and speech sounds (e.g., consonant-vowel pairs), then progresses through words, phrases, and sentences, culminating in natural conversation. Each level must be completed with at least 80% accuracy before proceeding to the next one.
  The structure is modeled after traditional voice therapies like resonant voice and aims to help participants succeed early and reduce mental fatigue. Daily homework includes seven short (2.5-minute) practice sessions, aligned with prior research showing this is a realistic and effective amount of practice.
  Arms: Hierarchical Conversation Training Therapy (CTT-H)
Other: Non Hierarchical method — The therapy includes four weekly sessions and several key techniques:
  Clear Speech: Speaking clearly, like leaving an important voicemail.
  Awareness Training: Paying attention to how the voice sounds and feels in the mouth and face.
  Negative Practice: Switching between their "bad" voice and "good" therapy voice to recognize and improve differences.
  Embedded Gestures: Briefly holding certain speech sounds to reduce vocal strain and boost clarity.
  Prosody and Projection: Working on pitch, rhythm, and speaking louder through better technique.
  Participants practice these skills throughout the day using a mobile app to track their progress and record a weekly sample. Unlike hierarchical models, components in CTT can be introduced in any order based on individual needs, making it flexible and personalized
  Arms: Non-Hierarchical Conversation Training Therapy (CTT)

SUMMARY:
This research study aims to evaluate the effect of treatment delivery method on voice outcomes over 12 months in people with a primary complaint of a voice problem, diagnosed with either non-phonotraumatic vocal hyperfunction, also known as primary muscle tension dysphonia (MTD) or phonotraumatic vocal hyperfunction, also known as benign vocal fold lesions (lesions).

The secondary objectives are:

* To evaluate acoustic correlates of clear speech and the relationship to vocal acoustic and patient-reported voice outcomes.
* To determine the association between overall dysphonia outcomes and adoption of clear speech.

DETAILED DESCRIPTION:
About 23 million Americans-roughly 1 in 13 people-suffer from voice problems at any given time. These issues can make it hard to speak clearly, lead to throat pain or fatigue, and affect daily life, work, and emotional well-being. The two most common types of voice problems are:

* Muscle tension dysphonia (MTD): when muscles in the throat are too tight during speaking.
* Benign vocal fold lesions: such as nodules or swelling on the vocal cords due to overuse or strain.

The most common treatment for these conditions is behavioral voice therapy, which involves working with a speech-language pathologist (SLP) to learn new ways to use the voice. However, over a third of patients drop out, and long-term success is uncertain. One major challenge is helping patients apply what they learn in therapy to their real-life conversations-a step often saved for the end of treatment or skipped entirely.

Traditional voice therapies often follow a strict step-by-step ("hierarchical") approach. Patients start with basic sounds or exercises and only work up to everyday speech later. But this method may not be the most effective, and many people struggle to use the new techniques outside the clinic.

To solve this problem, the research team developed a new method called Conversation Training Therapy (CTT). CTT flips the traditional approach: it begins with practicing clear, intentional speech in real conversation from the first session. This helps patients immediately apply new voice skills in real-life situations, which may lead to faster, more lasting results.

Studies have shown that CTT leads to meaningful improvements in voice-related quality of life both immediately and up to three months after therapy. It is now being used in national research studies and has gained recognition as a promising, evidence-based therapy. The current research will compare CTT to traditional methods over a full year, helping to answer important questions about what makes voice therapy work-and how to help more people benefit from it long-term.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Diagnosis of either primary muscle tension dysphonia of the hyperadducted type or benign vocal fold lesions.
* No neuro-laryngologic or age-related vocal fold changes (e.g., atrophy)
* No history of voice therapy or voice surgery in the last year
* No history of other serious chronic medical conditions that may affect voice (per patient report), Normal hearing (determined by pure tone audiometry), stimulable and appropriate for behavioral voice intervention as determined by a voice-specialized speech-language pathologist and laryngologist,
* Willingness to attend all therapeutic interventions and follow-up sessions
* Willingness to use a smartphone to record practice

Exclusion Criteria:

* History of voice therapy or voice surgery in the last year
* Serious chronic medical condition that may affect voice (per patient report)
* Abnormal hearing ability (despite appropriate amplification)
* Other laryngeal disorders not attributed to primary MTD and benign vocal fold lesions,
* Not stimulable or inappropriate for behavioral voice intervention as determined by a voice-specialized speech-language pathologist and laryngologist
* Unwillingness to attend therapeutic intervention and follow-up sessions
* Unwillingness to use a smartphone to record practice
* Pregnant women
* Prisoners
* Cognitive impairment or impaired decision-making capacity

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Change in Voice Handicap Index-10 (VHI-10) score | During intervention (4 week period of active treatment: Week 1, Week 2, Week 3, Week 4) immediately post treatment ( week 5), 3month, 6 month and 12-months post treatment
  The Voice Handicap Index-10 (VHI-10) is a 10-question survey used to measure how much a voice problem affects a person's daily life. Scores range from 0 to 40, with higher scores indicating a greater perceived voice handicap. Each item is rated from 0 ("never") to 4 ("always") A higher score means greater voice-related disability as perceived by the patient.
Change in vowel space | During intervention (4 week period of active treatment: Week 1, Week 2, Week 3, Week 4) immediately post treatment ( week 5), 3month, 6 month and 12-months post treatment.
  Change in vowel space refers to alterations in the acoustic range of vowel production-specifically, how far apart vowels are from each other in the formant frequency space (typically plotted as F1 vs F2, the first and second formants). It reflects the clarity, precision, and distinctiveness of vowel articulation during speech.
  Vowel space will be measured through acoustic analysis of participants' spoken sentences from the Sentence Intelligibility Test (SIT).
  These sentences include both corner vowels (e.g., heed, had, hod, who'd) and non-corner vowels (e.g., hid, head, hut, hood), allowing for detailed tracking of articulatory patterns

SECONDARY OUTCOMES:
Auditory- Perceptual severity | Baseline , 3 month, 6 month, 12 month
  It is measured using the CAPE-V (Consensus Auditory-Perceptual Evaluation of Voice) scale, a standardized tool.
  Raters (blinded speech-language pathologists) will score overall voice severity on a 0-100 mm visual analog scale-with 0 indicating no perceived disorder and 100 indicating extremely severe voice abnormality.
  This rating captures a listener's perception of qualities like roughness, breathiness, strain, and overall voice quality.
Stroboscopic changes: Glottal Closure | Baseline, Post intervention (1 week), 3 month, 6 month, 12 month
  Visual inspection during phonation. Described as: complete, anterior gap, posterior gap, hourglass, spindle, irregular, incomplete.
  Assessments will be made using a standardized tool called VALI (Voice-Vibratory Assessment with Laryngeal Imaging), which scores multiple vibratory features.
Stroboscopic changes: Amplitude | Baseline, Post intervention (1 week), 3 month, 6 month, 12 month
  Observed lateral movement of vocal folds. Subjectively rated as reduced, normal, or excessive. Assessments will be made using a standardized tool called VALI (Voice-Vibratory Assessment with Laryngeal Imaging), which scores multiple vibratory features.
Stroboscopic changes: Mucosal Wave | Baseline, Post intervention (1 week), 3 month, 6 month, 12 month
  Magnitude of mucosal membrane during vibration. Scored on a 0-10 scale based on visibility and extent Assessments will be made using a standardized tool called VALI (Voice-Vibratory Assessment with Laryngeal Imaging), which scores multiple vibratory features.
Stroboscopic changes: Free edge contour | Baseline, Post intervention (1 week), 3 month, 6 month, 12 month
  Shape of vocal fold edges during vibration. Rated as: normal, convex, concave, irregular, or rough Assessments will be made using a standardized tool called VALI (Voice-Vibratory Assessment with Laryngeal Imaging), which scores multiple vibratory features.
Stroboscopic changes: Phase closure | Baseline, Post intervention (1 week), 3 month, 6 month, 12 month
  Duration of open vs. closed phase during each vibratory cycle. Rated as: open phase dominates, equal, closed phase dominates Assessments will be made using a standardized tool called VALI (Voice-Vibratory Assessment with Laryngeal Imaging), which scores multiple vibratory features.
Stroboscopic changes: Phase symmetry | Baseline, Post intervention (1 week), 3 month, 6 month, 12 month
  Synchrony of left and right vocal fold movement. Rated as: symmetric or asymmetric Assessments will be made using a standardized tool called VALI (Voice-Vibratory Assessment with Laryngeal Imaging), which scores multiple vibratory features.
Stroboscopic changes: Regularity percentage | Baseline, Post intervention (1 week), 3 month, 6 month, 12 month
  Consistency of vibratory cycles over time. Expressed as % of time vibration is regular Assessments will be made using a standardized tool called VALI (Voice-Vibratory Assessment with Laryngeal Imaging), which scores multiple vibratory features.
Aerodynamic changes: Average airflow in speech | Baseline, Post intervention (1 week), 3 month, 6 month, 12 month
  Average airflow in speech - measures how much air passes through the vocal folds per second during phonation (typically in liters/second or mL/second). Abnormal airflow can indicate vocal fold dysfunction, such as incomplete closure or excessive strain.
  This data will be collected using the Phonatory Aerodynamic System 6600 (PAS) by PENTAX, a specialized tool for assessing voice aerodynamics. The PAS system uses a mask and microphone setup to capture airflow and sound pressure during structured speech tasks.
Aerodynamic changes: Average number of breaths | Baseline, Post intervention (1 week), 3 month, 6 month, 12 month
  Average number of breaths - counts how many breaths a speaker takes during a speech task. Higher breath counts may reflect inefficient voice use or reduced respiratory support.
  This data will be collected using the Phonatory Aerodynamic System 6600 (PAS) by PENTAX, a specialized tool for assessing voice aerodynamics. The PAS system uses a mask and microphone setup to capture airflow and sound pressure during structured speech tasks.
Aerodynamic changes: Average speaking duration | Baseline, Post intervention (1 week), 3 month, 6 month, 12 month
  Speaking duration is how long it takes the person to speak the entire passage. This data will be collected using the Phonatory Aerodynamic System 6600 (PAS) by PENTAX, a specialized tool for assessing voice aerodynamics. The PAS system uses a mask and microphone setup to capture airflow and sound pressure during structured speech tasks.
Adherence | Baseline, end of study (12 month)
  Practice will be analyzed for frequency of practice per week
Practice fidelity | Baseline, end of study (12 month)
  Practice fidelity will be assessed via analysis of audio-recordings for presence/absence of negative practice and type of practice (i.e. conversation, monology, recitation, reading aloud).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Gillespie, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Voice Center at Emory University Hospital Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will generate multi-modal data from 120 participants with voice disorders, including acoustic, aerodynamic, perceptual, and imaging data (\~30GB .wav/.nsp files; 135GB laryngeal videos), patient-reported outcomes (\~50MB REDCap exports), therapy session videos (\~2TB .mp4 files), and practice audio files. Core data (e.g., VHI-10 scores, voice outcomes) will be stored and shared via the Open Science Framework (OSF), adhering to NIH FAIR data principles. Files <3MB (e.g., protocols, VHI-10 raw data) may be included in publications as appendices.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Datasets will be uploaded to OSF within 6 months of their collection, beginning 4 months after the award begins
Access Criteria: Acoustic, aerodynamic, visual, and auditory perceptual and patient-reported outcomes data will be made available on the Open Science Framework Repository. This repository is an open-access, free platform designed for data preservation and sharing. De-identified datasets and metadata will be publicly accessible through this repository.
  PI will maintain up-to-date ORCID records with persistent unique identifiers such as DOIs for publications and funder IDs to assist findability. DOIs will be searchable in the Open Science Framework Repository.